CLINICAL TRIAL: NCT04392752
Title: Effects of the Fitness Competition Period on Body Composition, Neuromuscular Performance, Physiological and Psychological Factors in Fitness Athletes
Brief Title: Fitness Study 2020
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Jyvaskyla (Other)
Collaborators: Finnish Institute for Health and Welfare (Other Government)
Responsible Party: Principal Investigator, Ville Isola, Co-Investigator, University of Jyvaskyla
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: fitnessjyvaskyla
Record Dates: First submitted 2019-09-25; First posted 2020-05-19 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Weight Reduction; Diet; Deficiency
MeSH Terms: conditions — Weight Loss; Malnutrition

STUDY DESIGN:
Intervention Model Description: This study includes four laboratory testing sessions over the 50-week period. Testing sessions will be performed over one week. Time points include testing before the diet or the control period start (PRE), one week before the competition (MID), after the competition (COMP) and after a recovery period (POST), during which the participants are advised to continue their normal training regimen, but to stop competition dieting. Participants will spend three hours in the laboratory between 0700-1300. The control group will be advised to maintain their normal physical activity diet throughout the study. The participants will be given identification numbers and the research group is blinded so that they do not know which group participants belong to. All measurements will be conducted at the same time (always within max ±1 hour) due to the importance of standardizing the time of the day of measurements.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participants (Experimental): The participants are recruited via the University of Jyväskylä and Finnish Fitness Sports Association web page and social media channels. An online pre-study questionnaire are sent to randomly chosen athletes and control group candidates who claim to fulfill the inclusion criteria and volunteer for the study. The participants selected for the study filled an additional questionnaire which is subsequently reviewed by the physician of the study to confirm that they will meet inclusion criteria relating to health.
  Interventions: Other: Dieting intervention
- Control (No Intervention): The target is 15 male ja 15 female participants for both the control and intervention groups. To be included, participants need to be with two or more years of resistance training experience, similar to our previous study in females (Hulmi et al. 2017). If more than 15+15 control participants sign up for the study, the final group will be matched to the intervention group based on age, height, weight, and training experience reported on the pre-study questionnaire. The control group maintain their normal nutrition and training during the study.

INTERVENTIONS:
Other: Dieting intervention — This study includes four laboratory testing sessions over the 50-week period. Testing sessions will be performed over one week. Time points include testing before the diet or the control period start (PRE), one week before the competition (MID), after the competition (COMP) and after a recovery period (POST), during which the participants are advised to continue their normal training regimen, but to stop competition dieting. Participants will spend three hours in the laboratory between 0700-1300. The control group will be advised to maintain their normal physical activity diet throughout the study. The participants will be given identification numbers and the research group is blinded so that they do not know which group participants belong to. All measurements will be conducted at the same time (always within max ±1 hour) due to the importance of standardizing the time of the day of measurements.
  Arms: Participants

SUMMARY:
The experimental participant group (n=15+15) includes male and female fitness athletes during their ~25 week competition preparation in fall 2019 for the Finnish national championships. Participants must have at least two years of goal-oriented gym training and their health status will be determined before measurements via an online pre-study questionnaire. The control group (n=15+15) will maintain their normal training and diet without competing during the study period. Otherwise, the control group is matched with the athletic group based on age, height, weight and training experience. Participants selected for the study will complete an additional questionnaire to be reviewed by the study physician to confirm that participants meet the health status inclusion criteria. This study includes four laboratory testing sessions over the 50-week period. Time points include testing before the diet or the control period start (PRE), one week before the competition (MID), after the competition (COMP) and after a recovery period (POST). During COMP-POST the participants are advised to continue training, but to stop competition dieting."Measurements will include body composition (fat mass and fat free mass by bioimpedance, DXA and skinfolds), resting metabolic rate (indirect calorimetry), vastus lateralis and triceps brachii muscle-cross sectional area, subcutaneous fat thickness from ultrasonography and circulating hormone analysis. Also, whole blood will be analyzed for hemoglobin and hematocrit and systems biology approach: e.g. serum metabolome and possibly also other analysis. Lower body maximal voluntary isometric force will be measured via knee extension machine device. Average weekly physical activity will be determined with a wrist-worn uni-axial accelerometer. Training and dietary data (nutrient intake, volume, intensity etc.) will be collected via nutrition and training diaries. Psychological questionnaires will be conducted via an online survey.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the effects of competition preparation and recovery period on body composition, the endocrine system, metabolic rate, physical activity and performance, dietary and training habits and mood state in fitness athletes.

Metabolic and hormonal adaptations due to weight loss oppose further weight loss and pose challenges for maintaining reduced body weight. Fitness competition preparation (i.e., a substantial decrease in body fat mass without notable decreases in muscle mass) is accomplished by restricting total daily energy intake and increasing dosage of aerobic exercise dosage while maintaining high levels of resistance training and dietary protein. There is sparse research regarding the effects of the competition preparation and the recovery period afterwards the competition on body composition, neuromuscular performance, hormone balance, and metabolic rate. Additionally, the effects of preparation on mood states and on systems biology is not well studied.

The present study will help us understand the degree to which adaptations are due to the preparation and recovery process, or as a consequence of reaching the desired body composition (or some combination thereof). In turn, the findings may serve to help develop coaching guidelines for fitness athletes which minimize unfavorable adaptations to preparation and minimize the stress of the process. Participants will be notified of the research procedures, requirements, benefits and risks before providing written informed consent. The study will include one doctoral thesis and four scientific research articles during 2020-2024. Measurements of the study will be conducted during the spring of 2019 and 2020. Analyzing the results will occur during the year 2021 and the scientific publications will be reported by the end of 2024. The study is funded externally by the Finnish Fitness Sports Association and we will apply to additional, appropriate research grants. A large amount of data will be collected and processed which requires good management and leadership. In order to avoid risks, a comprehensive data management plan will be made for the study.

ELIGIBILITY:
Inclusion Criteria:

* two or more years of resistance training experience,
* participants must be 22-40 years old
* No 3 shiftwork
* Participants must be preparing for the Finnish Fitness Sports Association's national championships 2019 in the bodybuilding or men's or women´s divisions to be eligible intervention group.

Exclusion Criteria:

* diagnosed with chronic diseases
* prescribed medications
* using performance-enhancing drugs
* competing in the bodybuilding or men's fitness divisions autumn 2019 or 2020
* competing junior or master categories
* competing at non-drug tested competitions

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-02-02 (Actual); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in body composition during the competition preparation and after the recovery period | (-25 week, -1 week, +1-day, +25 week)
  Fat mass (kg) will be estimated by Dual-energy X-ray absorptiometry (DXA, Lunar Prodigy Advance, GE Medical Systems-Lunar, Madison WI USA) using methods similar to Hulmi et al. (2015; 2017) in a fasted state. The analysis (using enCORE 2005, version 9.30 and Advance 12.30) will provide total fat mass (kg). There will be 3 measurements.

SECONDARY OUTCOMES:
Change in physical performance during the competition preparation and after the recovery period | (-25 week, -1 week, +25 week)
  Maximal isometric force (Nm) output of the knee extensors of the right leg is assessed using an isokinetic dynamometer (Type 9287, Kistler, Switzerland connected to Spike 2™ software. There will be 3 measurements.
Change in physical activity and training diaries during the competition preparation and after the recovery period | -25-week, -20-wee, 16-week, -12-week, -8-week, -4-week, -1week, +1-week +4-week, +8-wee, +12-week, +16-week, +20-week, +25-week
  Mean weekly physical activity (MET) will be monitored using a wrist-worn uni-axial accelerometer Polar Active (Brugniaux et al. 2008). The participants are to wear the Polar Active continuously during a 3-week periods. The activity measurement last for 21 days. During the activity measurement, the wrist-worn accelerometer is worn at all times, except in sauna or bath. Polar Active uses sex, age, body mass, and height as an input to convert the measured acceleration signal to METs with the epoch length of 30 s. Polar Active has been found to correlate well (R2 = 0.74) with the doubly labeled water technique while assessing energy expenditure during a 7- day period of military training (Kinnunen et al., 2012). Data will be collect every month. There will be 14 measurements.
Change in resting metabolic rate during the competition preparation and after the recovery period | (-25 week, -1 week, +25 week)
  Resting metabolic rate (J/h·kg) will be measured with indirect calorimetry via respiratory quotient (RQ) assessments. Measurement is performed in a supine position over a 10-min period in a dark, thermos-neutral and quiet laboratory space. Expired gases during the tests are continuously analyzed over the 10 min period (Compher et al. 2006). There will be 3 measurements.
Change in different omics in during the competition preparation and after the recovery period | (-25 week, -1 week, +1-day, +25 week)
  A high-throughput serum Nuclear Magnetic Resonance (NMR) metabolomics platform will be used for the absolute quantification of serum lipids and metabolite profile. The NMR metabolome assay yields a total of 228 different metabolites, including an array of lipoprotein subclasses (e.g., VLDL, LDL, HDL), apolipoproteins, A-1 and B-100, serum free fatty acids, and a wide variety of small molecules such as glycolysis precursors, amino acids and inflammation biomarkers. In the platform, lipoproteins are divided into subclasses according to particle size. Serum metabolics will be quantified from acquired fasting blood samples by Brainshake (Finland) company, specializing in metabolomics quantification. Further, statistical analysis of provided data will be handled at Genomics and biomarkers unit, Institute for Health and Welfare (THL, Finland). There will be 4 measurements.
Chance in muscle subcutaneuous fat thickness in vastus lateralis muscle during the competition preparation and after the recovery period | (-25 week, -1 week, +1-day, +25 week)
  Vastus lateralis subcutaneous fat thickness (mm) will be examined (Hulmi et al. 2017) at the mid-thigh will be assessed using a B-mode axial plane ultrasound (model SSD-α10, Aloka, Tokyo, Japan) with a 10 MHz linear-array probe (60 mm width) in extended-ﬁeld-of-view mode (23 Hz sampling frequency). There will be 4 measurements.
Change in hormonal balance during the competition preparation and after the recovery period | (-25 week, -1 week, +1-day, +25 week)
  Free thyroxine (pmol/l) will be analyzed from serum with the Immunolite 2000 XPi, immunoassay system (Seimen Healtineers, Erlangen Germany).There will be 4 measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Juha P Ahtiainen, PhD, Study Director — Faculty od Sport and Health Sciences, University of Jyväskylä, Finland
Locations (1):
- University of Jyväskylä, Jyväskylä, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hulmi JJ, Isola V, Suonpaa M, Jarvinen NJ, Kokkonen M, Wennerstrom A, Nyman K, Perola M, Ahtiainen JP, Hakkinen K. The Effects of Intensive Weight Reduction on Body Composition and Serum Hormones in Female Fitness Competitors. Front Physiol. 2017 Jan 10;7:689. doi: 10.3389/fphys.2016.00689. eCollection 2016. PMID 28119632
- [Derived] Mikkonen R, Hackney AC, Hulmi J, Isola V, Ahtiainen J, Ihalainen J. Hormone Profiles After Planned Low Energy Availability Exposure in Naturally Menstruating and Hormonal Contraceptive Using Physique Athletes. Eur J Sport Sci. 2025 Dec;25(12):e70076. doi: 10.1002/ejsc.70076. PMID 41235908
- [Derived] Isola V, Hulmi JJ, Petaja P, Helms ER, Karppinen JE, Ahtiainen JP. Weight loss induces changes in adaptive thermogenesis in female and male physique athletes. Appl Physiol Nutr Metab. 2023 Apr 1;48(4):307-320. doi: 10.1139/apnm-2022-0372. Epub 2023 Jan 16. PMID 36645885